CLINICAL TRIAL: NCT06942572
Title: A Phase 1/2, First-in-Human, Open-label, Assessor-Masked, Randomized, Controlled, Dose Escalation/Expansion Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of a Subretinal Injection of SB-007 in Subjects With Stargardt Disease (STGD1) Caused by Bi-Allelic Autosomal Recessive Mutations in the ATP Binding Cassette Subfamily A Member 4 (ABCA4) Gene
Brief Title: A Phase 1/2, First-in-Human Dose Escalation/Expansion Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of a Subretinal Injection of SB-007 in Subjects With Stargardt Disease (STGD1)
Acronym: ASTRA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Splice Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB-007 CS-101; 2024-519535-42 (EudraCT Number)
Record Dates: First submitted 2025-02-18; First posted 2025-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stargardt Disease; Stargardt Macular Degeneration; Stargardt Macular Dystrophy
Keywords: Gene Therapy; SB-007; Splicebio; Stargardt; Stargardts Disease; SGDT1
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Intervention Model Description: Non-Randomised Dose Escalation (Part A) followed by Randomised Dose Expansion (Part B).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Non-Randomised Dose Escalation (Part A) is fully unmasked. Randomised Dose Expansion Cohort (Part B) masked to Study Dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 1 Dose Escalation - Low Dose (Experimental): Low Dose: Subjects will receive subretinal injection of SB-007 in the low dose group
  Interventions: Genetic: SB-007
- Phase 1 Dose Escalation - Medium Dose (Experimental): Medium Dose: Subjects will receive subretinal injection of SB-007 in the medium dose group
  Interventions: Genetic: SB-007
- Phase 1 Dose Escalation - High Dose (Experimental): High Dose: Subjects will receive subretinal injection of SB-007 in the high dose group
  Interventions: Genetic: SB-007
- Phase 2 Dose Expansion: Dose 1 from Phase 1 Randomised Arm (Experimental): Subjects will receive a subretinal injection of SB-007 with Maximum tolerated dose (MTD) from Phase 1
  Interventions: Genetic: SB-007
- Phase 2 Dose Expansion: Dose 2 from Phase 1 Randomised Arm (Experimental): Subjects will receive a subretinal injection of SB-007 with lower dose than Maximum tolerated dose (MTD) from Phase 1
  Interventions: Genetic: SB-007
- Phase 2 No Intervention - Randomised Control Arm (No Intervention): No Intervention Control Arm: Subject will not receive any active study intervention

INTERVENTIONS:
Genetic: SB-007 — Subretinal Administration of SB-007
  Arms: Phase 1 Dose Escalation - High Dose; Phase 1 Dose Escalation - Low Dose; Phase 1 Dose Escalation - Medium Dose; Phase 2 Dose Expansion: Dose 1 from Phase 1 Randomised Arm; Phase 2 Dose Expansion: Dose 2 from Phase 1 Randomised Arm

SUMMARY:
This Phase 1/2 study will evaluate the safety, tolerability, and preliminary efficacy of subretinal SB-007 administration to determine dose selection in subjects with Stargardt's Type 1 (STGD1).

This is a multicenter study which will enroll approximately 57 subjects, followed up over a 96 week period post treatment after a single administration of SB-007.

DETAILED DESCRIPTION:
Inherited retinal dystrophies (IRDs) are a group of genetically and clinically heterogeneous disorders caused by progressive degeneration of photoreceptor (PR) rods, cones, or both. The majority of IRDs are characterized by retinal degeneration, which can lead to significant vision impairment and blindness and are thus serious and debilitating conditions. Most IRDs have no treatment options.

Stargardt disease (STGD1) is an autosomal recessive IRD that generally manifests during childhood or early adulthood. It has an estimated prevalence of 1 in 8,000 to 10,000 patients. STGD1 is due to mutations in the adenosine triphosphate (ATP)-binding cassette, sub-family A, member 4 (ABCA4) gene. The ABCA4 protein is an ATP-binding cassette (ABC) transporter expressed in PR outer segments in both rods and cones. This protein plays a critical role in the visual phototransduction cycle. Mutations in the ABCA4 gene adversely affect the metabolism of vitamin A, leading to deposition and build-up of lipofuscin containing bisretinoid toxins, such as N-retinylidene-N-retinylethanolamine (A2E), in the PRs and retinal pigment epithelium (RPE) cells. This accumulation of lipofuscin causes the formation of yellowish flecks over the macula and toxins such as A2E lead to oxidative stress and death of RPE cells and light-sensing photoreceptors.

Gene therapies are emerging as potentially viable treatments for a variety of IRDs. Many of these therapies are based on the use of adeno-associated virus (AAV) vectors containing DNA that encodes a functional gene to replace a defective gene.

Although AAV vectors have good biological characteristics (i.e., high transduction efficiency, genetic stability) and acceptable safety profiles (non-immunogenic, non-pathogenic, few serious adverse effects), one drawback is its packaging capability. Until recently, use of AAV vectors was not considered appropriate for STGD1 gene therapies since the ABCA4 gene is too large and exceeds the capacity of AAV vectors. However, SpliceBio, a genetic medicines company, has developed a proprietary protein splicing intein platform using dual AAV vectors that enables the delivery of genes too large for conventional AAV vector systems. SpliceBio is using this technology to develop a genetic treatment for STGD1.

SB-007 is a new gene therapy investigational medicinal product based on dual AAV8 gene delivery for the full-length reconstitution of the ABCA4 protein inside the target cell using protein trans-splicing mediated by small polypeptidic proprietary sequences called split-inteins. While each alone are inactive, the co-expression of the 2 vectors is expected to lead to highly efficient PTS and reconstitution of the full-length biologically active ABCA4 protein in target photoreceptor cells. Further, SB-007 is anticipated to enable long-term expression of a functional wild type ABCA4 protein in the retina of patients and thus slow or blunt further vision loss after a single subretinal administration.

First-in-human trials are conducted primarily to determine the safe dose range for further clinical development of promising drug candidates. This first-in-human study is being conducted to identify doses of SB-007 that are safe and demonstrate a potential efficacy signal in subjects with moderate or advanced STGD1.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study participation, subjects must meet the following criteria:

1. Provide written consent. Subjects under legal age will also provide informed assent according to guidelines set forth by the same.
2. Are male or female adolescents and adults, aged as follows:

   1. In Part A, subjects will be ≥18 to ≤65* years (inclusive)
   2. In Part B, subject age is planned as ≥12 to ≤65* years (inclusive) *Subjects aged >65 years may be eligible in Parts A and B, following discussion with, and approval by, the Medical Monitor.
3. Are able to understand and comply with the study procedures.
4. Have a diagnosis of STGD1 caused by bi-allelic pathogenic, or likely pathogenic, variants in the ABCA4 gene confirmed genotypically by an accredited genetic testing laboratory
5. Clinical evidence consistent with Stargardt Disease type 1.
6. For women of child-bearing potential (WOCBP), have a negative pregnancy test at Screening and, if due to receive active treatment, at Day 0.
7. For both WOCBP and male subjects (or their female partners who are of child-bearing potential), agree to either strict abstinence or, if sexually active, use an acceptable contraception measure for 3 months from Day 0
8. Must have clear ocular media and adequate pupillary dilation in the study eye, including no allergy to dilating eyedrops, to permit good quality retinal imaging.
9. Fulfil visual acuity criteria based on ETDRS letter chart
10. Fulfil baseline lesion size measurement, as measured by the Reading Center
11. Evidence of disease progression as determined by the Medical Monitor following consultation with the Investigator.

Exclusion Criteria:

Subjects must be excluded from participating in the study if they:

1. Have had any intraocular surgery (including cataract surgery) or thermal laser within 90 days of the Screening Visit or planned intraocular surgery (including cataract surgery) or thermal laser during the period of the study, in the study eye.
2. Have had any major surgical procedure within 30 days of the Screening Visit or planned or anticipated major surgery during the period of the study.
3. Have two pathogenic or likely pathogenic variants in IRD genes (other than ABCA4) or a single pathogenic or likely pathogenic variant in autosomal dominant or X-linked IRD genes.
4. Have a history of amblyopia in the study eye.
5. Are unwilling to stop taking the following products at Screening and throughout the study:

   1. Supplements containing vitamin A or beta-carotene, liver-based products.
   2. Prescription oral retinoids. Topical products containing vitamin A or retinoids are not exclusionary.
6. Have any ophthalmic history of gene therapy, stem cell therapy, surgical implantation of prosthetic retinal chips, or intravitreal or sub-retinal or supra-choroidal injections.
7. Have received any investigational therapy within 90 days of the Screening Visit or 5 half-lives, whichever is longer.
8. Have known serious allergies to the fluorescein dye that might be used to measure IOP, ocular dilating drops, topical ocular anesthetic, steroid medication, or components of the SB-007 formulation.
9. Have any significant ocular or non-ocular disease/disorder which, in the opinion of the Investigator and with concurrence of the Medical Monitor, may either put the subject at risk because of participation in the study, may influence the results of the study, or affect the subject's ability to participate in the study.
10. Are an immediate family member (e.g., child, sibling) of the Sponsor or study site personnel.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Measures | 96 weeks
  Safety and tolerability assessed by incidence and/or clinically significant changes in ocular and non-ocular AEs

SECONDARY OUTCOMES:
Efficacy Measure: Change from baseline in lesion size using autofluorescence (FAF) | 96 weeks (Screening to 96 weeks post SB-007 administration)
  Change from baseline in lesion size growth (mm^2) on FAF imaging compared between SB-007 and untreated control at Week 96, adjudicated by a Central Reading Center
Other Efficacy Measure: Change from baseline in retinal sensitivity | 48 and 96 weeks (Screening to 48 and 96 weeks post SB-007 administration)
  Change from baseline in retinal sensitivity based on microperimetry at Weeks 48 and 96
Other Efficacy Measure: Change from baseline in BCVA (Best Corrected Visual Acuity) | 48 and 96 weeks (Screening to 48 and 96 weeks post SB-007 administration)
  Change from baseline in BCVA using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score at Weeks 48 and 96
Other Efficacy Measure: Change from baseline in LLVA (Low Luminance Visual Acuity) | 48 and 96 weeks (Screening to 48 and 96 weeks post SB-007 administration)
  Change from baseline in LLVA using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at Weeks 48 and 96. A higher score represents better vision at low light levels.
Other Efficacy Measure: Change in Quality of Life measure using MRDQ | 48 and 96 weeks (Screening to 48 and 96 weeks post SB-007 administration)
  The Michigan Retinal Dystrophy Questionnaire (MRDQ) is a patient reported outcome measure that will be administered to assess visual function in subjects with Inherited Retinal Dystrophies
Other Efficacy Measure: Change in Quality of Life measure using PGI questionnaires | 48 and 96 weeks (Screening to 48 and 96 weeks post SB-007 administration)
  These Patient Global Impression (PGI) scales evaluate all aspects of a patients health and assesses if there has been an improvement or decline in clinical status

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCHealth Sue Anschutz-Rodgers Eye Center,, Aurora, Colorado
  - Bascom Palmer Eye Institute, Miami, Florida
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Oregon Health & Science University, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: SpliceBio Website — https://splice.bio/clinical/